CLINICAL TRIAL: NCT05803122
Title: Validation of the I-UDS Neuropsychological Battery in Patients With Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Validation of the I-UDS Neuropsychological Battery
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: IRCCS Associazione Oasi Maria SS. ONLUS, Troina, Italy (Unknown); IRCCS Istituto Auxologico Italiano, Milano, Italy (Unknown); Fondazione IRCCS Istituto Neurologico Carlo Besta, Milano, Italy (Unknown); IRCCS San Raffaele (Other); Fondazione IRCCS Santa Lucia, Roma, Italy (Unknown); IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Milano, Italy (Unknown); IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy (Unknown); IRCCS Don Gnocchi, Milano, Italy (Unknown); IRCCS Ospedale Maggiore Policlinico, Milano, Italy (Unknown); IRCCS AOU San Martino, Genova, Italy (Unknown); IRCCS SDN, Napoli, Italy (Unknown); IRCCS Fondazione Salvatore Maugeri, Pavia, Italy (Unknown); IRCCS Istituto delle Scienze Neurologiche di Bologna (Other); Istituto Di Ricerche Farmacologiche Mario Negri (Other); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other)
Responsible Party: Sponsor
Other Study IDs: I-UDS2022
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
Keywords: Neuropsychological tests; UDS; Alzheimer's Disease; Mild Cognitive Impairment; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Mild Cognitive Impairment (MCI): Patients with diagnosis of MCI based on diagnostic research criteria , after a protocol of clinical, neuropsychological, structural brain imaging evaluation and biomarkers positivity assessment (amyloid-Positron Emission Tomography (PET) and/or Cerebral Spinal Fluid -CSF).
  Interventions: Other: Uniform Data Set (UDS) neuropsychological battery
- Patients with Alzheimer's Disease (AD): Patients with diagnosis of AD based on diagnostic research criteria , after a protocol of clinical, neuropsychological, structural brain imaging evaluation and biomarkers positivity assessment (amyloid-PET and/or CSF).
  Interventions: Other: Uniform Data Set (UDS) neuropsychological battery

INTERVENTIONS:
Other: Uniform Data Set (UDS) neuropsychological battery — Uniform Data Set (UDS) neuropsychological battery was administered to patients with Mild Cognitive Impairment (MCI) and patients with Alzheimer's Disease

SUMMARY:
The current project entails the validation of the Italian version of the Uniform Data Set (I-UDS) neuropsychological in patients with neurodegenerative diseases, specifically in patients with Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD). Specifically, the final aim is to explore the ability of the battery to differentiate the cognitive profiles of the two groups of patients.

DETAILED DESCRIPTION:
The harmonization of procedures for neuropsychological assessment in dementia disorders is essential for the development of shared activities and projects within the IRCCS Network of Neuroscience and Neurorehabilitation (RIN). To this end, a previous project of the network was dedicated to the translation and adaptation of the Uniform Data Set (UDS) neuropsychological battery, following the similar initiative of the National Alzheimer's Coordinating Center (NACC) USA . This project led to the creation of the I-UDS, which can be administered via a tablet application and consists of tests aimed at investigating different cognitive domains, namely memory, attention, language, executive and visuospatial skills. Normative data were obtained from a sample of 433 healthy participants. In order to be able to use the I-UDS battery in clinical and research settings, it is essential to validate its application in patients with neurodegenerative diseases. In particular, in line with the NACC initiative, the battery aims to trace and highlight the continuum between Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD). The present multicenter study therefore aims to test the I-UDS battery in patients with clinical diagnoses of MCI and AD, in order to explore its ability to differentiate the cognitive profiles of the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MCI or AD based on diagnostic research criteria after a protocol of clinical, neuropsychological, structural brain imaging evaluation and biomarkers positivity assessment (amyloid-PET and/or CSF);
* performance in the Mini-Mental State Examination (MMSE) above/equal 20 (score corrected for age and education);

Exclusion Criteria:

* prior/current cerebrovascular disorders;
* a history of traumatic brain injury, brain tumors, stroke;
* concomitant medical, sensory and/or motor deficits possibly affecting performance;
* a history of alcohol and/or drug abuse;
* use of medications influencing cognitive functions.

Ages: 40 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be administered the neuropsychological battery of the Italian Uniform Data Set (I-UDS) through a dedicated tablet application, and consisting of tests aimed at investigating the main cognitive domains, i.e. memory, attention, language, executive and visual-spatial skills. The duration of battery administration is approximately 45 minutes.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
I-UDS battery | One time
  Patients' scores in the tests of the I-UDS battery

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cappa, MD, Principal Investigator — Dementia Research Center
Locations (1):
- Dementia Research Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] McKhann GM, Knopman DS, Chertkow H, Hyman BT, Jack CR Jr, Kawas CH, Klunk WE, Koroshetz WJ, Manly JJ, Mayeux R, Mohs RC, Morris JC, Rossor MN, Scheltens P, Carrillo MC, Thies B, Weintraub S, Phelps CH. The diagnosis of dementia due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):263-9. doi: 10.1016/j.jalz.2011.03.005. Epub 2011 Apr 21. PMID 21514250
- [Background] Weintraub S, Besser L, Dodge HH, Teylan M, Ferris S, Goldstein FC, Giordani B, Kramer J, Loewenstein D, Marson D, Mungas D, Salmon D, Welsh-Bohmer K, Zhou XH, Shirk SD, Atri A, Kukull WA, Phelps C, Morris JC. Version 3 of the Alzheimer Disease Centers' Neuropsychological Test Battery in the Uniform Data Set (UDS). Alzheimer Dis Assoc Disord. 2018 Jan-Mar;32(1):10-17. doi: 10.1097/WAD.0000000000000223. PMID 29240561
- [Background] Weintraub S, Salmon D, Mercaldo N, Ferris S, Graff-Radford NR, Chui H, Cummings J, DeCarli C, Foster NL, Galasko D, Peskind E, Dietrich W, Beekly DL, Kukull WA, Morris JC. The Alzheimer's Disease Centers' Uniform Data Set (UDS): the neuropsychologic test battery. Alzheimer Dis Assoc Disord. 2009 Apr-Jun;23(2):91-101. doi: 10.1097/WAD.0b013e318191c7dd. PMID 19474567
- [Result] Conca F, Esposito V, Rundo F, Quaranta D, Muscio C, Manenti R, Caruso G, Lucca U, Galbussera AA, Di Tella S, Baglio F, L'Abbate F, Canu E, Catania V, Filippi M, Mattavelli G, Poletti B, Silani V, Lodi R, De Matteis M, Stanzani Maserati M, Arighi A, Rotondo E, Tanzilli A, Pace A, Garramone F, Cavaliere C, Pardini M, Rizzetto C, Sorbi S, Perri R, Tiraboschi P, Canessa N, Cotelli M, Ferri R, Weintraub S, Marra C, Tagliavini F, Catricala E, Cappa SF. Italian adaptation of the Uniform Data Set Neuropsychological Test Battery (I-UDSNB 1.0): development and normative data. Alzheimers Res Ther. 2022 Aug 19;14(1):113. doi: 10.1186/s13195-022-01056-x. PMID 35982477